CLINICAL TRIAL: NCT03592173
Title: Non-Invasive Stimulation for Improving Motor Function in Spinal Cord Injury
Brief Title: Non-Invasive Stimulation for Improving Motor Function
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kathleen Friel (Other)
Collaborators: Burke Medical Research Institute (Other)
Responsible Party: Sponsor-Investigator, Kathleen Friel, Laboratory Director, Burke Medical Research Institute
Organization: Burke Medical Research Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BRC391
Record Dates: First submitted 2018-05-16; First posted 2018-07-19 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Thirty chronic SCI participants will given the SAS intervention and a control intervention in a randomized cross-over study, with at least one week between interventions. Each patient will be required to attend the Burke Medical Research Institute on three occasions. We will use a within-subjects design, to test changes in neurophysiologic and voluntary measures after intervention with respect to baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- SAS20 (Experimental): The paired stimulation (SAS) will be comprised of patient adjusted subthreshold TMS (80% of resting motor threshold over optimal site for soleus muscle), delivered 20ms prior to a peripheral nerve stimulus in the popliteal fossa and will be repeated at 0.1 Hz for 15 minutes (90 stimuli pairs).
  Interventions: Diagnostic Test: Paired TMS & Peripheral Nerve Stimulation
- SAS0 (Active Comparator): The paired stimulation (SAS) will be comprised of patient adjusted subthreshold TMS (80% of resting motor threshold over optimal site for soleus muscle), delivered 0ms prior to a peripheral nerve stimulus in the popliteal fossa and will be repeated at 0.1 Hz for 15 minutes (90 stimuli pairs).
  Interventions: Diagnostic Test: Paired TMS & Peripheral Nerve Stimulation
- SAS50 (Active Comparator): The paired stimulation (SAS) will be comprised of patient adjusted subthreshold TMS (80% of resting motor threshold over optimal site for soleus muscle), delivered 50ms prior to a peripheral nerve stimulus in the popliteal fossa and will be repeated at 0.1 Hz for 15 minutes (90 stimuli pairs).
  Interventions: Diagnostic Test: Paired TMS & Peripheral Nerve Stimulation

INTERVENTIONS:
Diagnostic Test: Paired TMS & Peripheral Nerve Stimulation — Method of assessing neurophysiology and activity of the spinal cord

SUMMARY:
The purpose of this study is to determine if spinal excitability is increased with a Spinal Associative Stimulation (SAS) protocol, and to determine the functional consequences of this technique on motor recovery.

DETAILED DESCRIPTION:
Recovery of motor function continues to be a problem following Spinal Cord Injury. Non-invasive brain stimulation techniques, targeting cortical areas, have been shown to enhance the excitability in the human motor cortex, and these changes in the motor cortex may be of significance for the rehabilitation of brain injured patients. However, little is known about the adaptational changes in the excitability/plasticity of spinal neural circuits in spinal cord injury patients.

The purpose of this study is to investigate the excitability of cortical and spinal inhibitory and excitatory mechanisms before and following a period of repetitive and synchronized dual peripheral nerve and brain stimulation. Repetitive, paired brain and peripheral nerve stimulation as a neuromodulatory tool, paired associative stimulation (PAS), has been well described. In this technique, stimuli are timed such that afferent and efferent volleys interact at the level of the cortex, that lead to a temporary enhancement of Motor Evoked Potential (MEP) amplitude in target muscles, and when applied repeatedly, lead to a sustained effect, outlasting the intervention period. This repetitive technique has been done in healthy subjects and patients with neurological diseases. By modifying the time between paired stimuli, the investigators will generate afferent/efferent interactions in the spinal cord.

The working hypothesis of this study is that the acute facilitation of the H-reflex during Paired TMS and peripheral nerve stimulation, may be harnessed to modulate spinal excitability (sustained increase in the MEP amplitude). That is, the investigators will test if similar to PAS, a change in excitability outlasting the stimulation/intervention period may occur with afferent/efferent interactions, although at the level of the spinal cord rather than the cortex, and be useful to strengthen residual pathways after damage to the spinal cord.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury subjects with chronic lesions (> 6 months after the injury)
* Motor incomplete lesion, measured by the American Spinal cord Injury Association (ASIA) Impairment Scale (AIS)
* Traumatic cause of lesion; d) Some degree of motor function in the ankle flexor and extensors (Low extremity Motor Score - LEMS≥3).

Exclusion Criteria:

* Motor and sensory complete lesion (AIS A); LEMS < 3;
* Non-traumatic cause of lesion
* Medically unstable condition
* Other concurrent neurological illness
* Presence of a potential TMS risk factor (detailed below)

Potential TMS risk factor:

* Damaged skin at the site of stimulation
* Presence of an electrically, magnetically or mechanically activated implant
* An intracerebral vascular clip, or any other electrically sensitive support system
* Metal in any part of the body, including metal injury to the eye
* A history of medication-resistant epilepsy in the family
* Past history of seizures or unexplained spells of loss of consciousness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-07 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in H-Reflex Threshold | Baseline compared with immediately after intervention
  Assessment of muscle reaction after stimulation of sensory fibers

SECONDARY OUTCOMES:
Lower Extremity Motor Score (LEMS) | Baseline, immediately after intervention
  Assessment of lower extremity strength in key muscles; maximal score of 50 with 20 or less indicating participant likely has limited ambulation.
Walking Index for Spinal Cord Injury (WISCI II) | Baseline, immediately after intervention
  This is a functional capacity scale that rank orders ambulation in people with spinal cord injury, by evaluating the amount of physical assistance, braces or devices required to walk 10 meters. Rank scores range from 0-20. A higher score is indicative of more independent ambulation.
10 Meter Walk Test | Baseline, immediately after intervention
  Measure of gait speed
Spinal Cord Independence Measure, Version 3 (SCIM III) | Baseline, immediately after intervention
  A disability rating scale developed to specifically address the ability of SCI patients to perform basic activities of daily living independently (including self-care, mobility, respiration and sphincter management)
Muscle Force | Baseline, immediately after intervention
  Amount of force recorded during maximal voluntary isometric contraction of a grip movement, recorded with a grip strength measurement device.
Anklebot | Baseline, immediately after intervention
  Lower extremity robotic device that provides kinematic evaluation data

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Friel, PhD, Study Director — Burke Medical Research Institute
Locations (1):
- Burke Medical Research Institute, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers at this time.

REFERENCES:
- [Background] Pascual-Leone A. Disrupting the brain to guide plasticity and improve behavior. Prog Brain Res. 2006;157:315-329. doi: 10.1016/s0079-6123(06)57019-0. PMID 17167918
- [Background] Deletis V, Schild JH, Beric A, Dimitrijevic MR. Facilitation of motor evoked potentials by somatosensory afferent stimulation. Electroencephalogr Clin Neurophysiol. 1992 Oct;85(5):302-10. doi: 10.1016/0168-5597(92)90106-l. PMID 1385090
- [Background] Hiersemenzel LP, Curt A, Dietz V. From spinal shock to spasticity: neuronal adaptations to a spinal cord injury. Neurology. 2000 Apr 25;54(8):1574-82. doi: 10.1212/wnl.54.8.1574. PMID 10762496
- [Background] Kumru H, Vidal J, Kofler M, Benito J, Garcia A, Valls-Sole J. Exaggerated auditory startle responses in patients with spinal cord injury. J Neurol. 2008 May;255(5):703-9. doi: 10.1007/s00415-008-0780-3. Epub 2008 Feb 21. PMID 18286318
- [Background] Rothwell JC. Techniques and mechanisms of action of transcranial stimulation of the human motor cortex. J Neurosci Methods. 1997 Jun 27;74(2):113-22. doi: 10.1016/s0165-0270(97)02242-5. PMID 9219881
- [Background] Kofler M, Valls-Sole J, Fuhr P, Schindler C, Zaccaria BR, Saltuari L. Sensory modulation of voluntary and TMS-induced activation in hand muscles. Exp Brain Res. 2008 Jul;188(3):399-409. doi: 10.1007/s00221-008-1372-2. Epub 2008 Apr 18. PMID 18421450
- [Background] Pascual-Leone A, Tarazona F, Keenan J, Tormos JM, Hamilton R, Catala MD. Transcranial magnetic stimulation and neuroplasticity. Neuropsychologia. 1999 Feb;37(2):207-17. doi: 10.1016/s0028-3932(98)00095-5. PMID 10080378
- [Background] Serranova T, Valls-Sole J, Munoz E, Genis D, Jech R, Seeman P. Abnormal corticospinal tract modulation of the soleus H reflex in patients with pure spastic paraparesis. Neurosci Lett. 2008 May 23;437(1):15-9. doi: 10.1016/j.neulet.2008.03.068. Epub 2008 Mar 28. PMID 18434014
- [Background] Boorman G, Becker WJ, Morrice BL, Lee RG. Modulation of the soleus H-reflex during pedalling in normal humans and in patients with spinal spasticity. J Neurol Neurosurg Psychiatry. 1992 Dec;55(12):1150-6. doi: 10.1136/jnnp.55.12.1150. PMID 1479394
- [Background] Poon DE, Roy FD, Gorassini MA, Stein RB. Interaction of paired cortical and peripheral nerve stimulation on human motor neurons. Exp Brain Res. 2008 Jun;188(1):13-21. doi: 10.1007/s00221-008-1334-8. Epub 2008 Mar 11. PMID 18330548
- [Background] Stefan K, Kunesch E, Benecke R, Cohen LG, Classen J. Mechanisms of enhancement of human motor cortex excitability induced by interventional paired associative stimulation. J Physiol. 2002 Sep 1;543(Pt 2):699-708. doi: 10.1113/jphysiol.2002.023317. PMID 12205201
- [Background] Ridding MC, McKay DR, Thompson PD, Miles TS. Changes in corticomotor representations induced by prolonged peripheral nerve stimulation in humans. Clin Neurophysiol. 2001 Aug;112(8):1461-9. doi: 10.1016/s1388-2457(01)00592-2. PMID 11459686
- [Background] Valls-Sole J, Alvarez R, Tolosa ES. Responses of the soleus muscle to transcranial magnetic stimulation. Electroencephalogr Clin Neurophysiol. 1994 Dec;93(6):421-7. doi: 10.1016/0168-5597(94)90148-1. PMID 7529691
- [Background] Hoffken O, Veit M, Knossalla F, Lissek S, Bliem B, Ragert P, Dinse HR, Tegenthoff M. Sustained increase of somatosensory cortex excitability by tactile coactivation studied by paired median nerve stimulation in humans correlates with perceptual gain. J Physiol. 2007 Oct 15;584(Pt 2):463-71. doi: 10.1113/jphysiol.2007.140079. Epub 2007 Aug 16. PMID 17702814